CLINICAL TRIAL: NCT02881151
Title: CT-DBS for Traumatic Brain Injury Using the Medtronic Activa PC+S System
Brief Title: Deep Brain Stimulation for the Treatment of Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaimie M. Henderson (Other)
Collaborators: Weill Medical College of Cornell University (Other); University of Utah (Other); Harvard Medical School (HMS and HSDM) (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Jaimie M. Henderson, John and Jene Blume - Robert and Ruth Halperin Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 37280
Record Dates: First submitted 2016-08-22; First posted 2016-08-26 (Estimated); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-11

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: Deep brain stimulation; DBS; Central thalamus; TBI; Traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Experimental): Subjects will be treated with deep brain stimulation throughout the study, with the exception of a brief, 21 day blinded withdrawal phase that will be undertaken to assess for any possible therapeutic effect.
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — Delivery of continuous, low-voltage electrical pulses to deep portions of the brain via an implantable pacemaker-like device.
  Other Names: DBS; CT-DBS; Central Thalamic DBS

SUMMARY:
This study involves the treatment of cognitive impairment secondary to moderate to severe brain injury using central thalamic deep brain stimulation. Although all patients will receive stimulation continuously through a surgically implanted pacemaker-like device, half of the patients will have the device deactivated during a blinded assessment phase. The device will be reactivated following this assessment and patients will have the option to continue stimulation in an open-label continuation.

DETAILED DESCRIPTION:
This preliminary safety study evaluates the use of the Medtronic Activa PC+S system and Medtronic Nexus-E system for central thalamic deep brain stimulation (CT-DBS) in the treatment of cognitive impairment secondary to traumatic brain injury (TBI). It involves a neurosurgical procedure in which electrodes are implanted in the brain, connected to an implanted pacemaker-like device in the chest. The proposed study, if successful, will provide supporting evidence for the development of a novel therapeutic approach utilizing CT-DBS to improve these enduring cognitive impairments arising in persons with multi-focal structural brain injuries. This research will address the critical gap of the lack of any available treatments. CT-DBS targets well-defined neuronal populations within the central thalamus that have known anatomical and physiological specializations, which not only provide a key role in arousal regulation during cognitively-mediated behaviors, but also exhibit a particular vulnerability to dysfunction in the setting of multi-focal, non-selective brain injuries.

Our proposed study aims to support development of CT-DBS as a novel therapeutic avenue for accessing cognitive reserve in patients with acquired brain injuries. In the proposed feasibility study of 6 subjects at a single investigational site, we will test the safety of CT-DBS in the severe traumatic brain injury (STBI) population with GOSE 6-7 level recovery and collect data to establish the translation of preclinical studies into human application of CT-DBS.

ELIGIBILITY:
Inclusion Criteria:

* History of moderate to severe TBI based on worst GCS score within first 48 hours of injury (acceptable GCS range = 3-12)
* Age 22-60
* At least 24 months from date of onset
* Fluent in English and able to independently provide consent
* Rating of upper moderate disability to lower good recovery on the Glasgow Outcome Scale-Extended (GOSE) at time of enrollment (acceptable GOSE range 5-7)
* Failure to return to pre-injury level of vocational or educational function
* Either receiving no CNS stimulants or other medications known to affect cognitive function, or on stable doses of these medications for the last three months

Exclusion Criteria:

* History of major developmental, neurologic, psychiatric or substance use disorder with evidence of disability prior to onset of TBI
* Major medical co-morbidities including: end stage renal failure, severe heart failure, coagulopathy, severe respiratory problems, severe liver failure, uncontrolled hypertension or other significant medical co morbidities
* Have had a documented seizure within 3 months of study screening (subjects may re-screen if seizure free after initial screen failure)
* Malignancy with < 5 years life expectancy
* Untreated / uncontrolled (severe at the time of enrollment) depression or other psychiatric disorder
* Women of childbearing age who do not regularly use an accepted contraceptive method
* Inability to stop anticoagulation therapy or platelet anti-aggregation therapy before, during and after surgery
* Previous DBS or other brain implants
* Previous ablative intracranial surgery
* Implantable hardware not compatible with MRI
* Condition requiring diathermy after DBS implantation
* Hardware, lesions or other factors limiting placement of electrodes in optimal target location in the judgment of the operating surgeon
* Concurrent enrollment in any other clinical trial
* Any condition or finding that, in the judgment of the PI, significantly increases risk or significantly reduces the likelihood of benefit from DBS

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaimie M Henderson, MD, Study Director — Stanford University
Locations (1):
- Stanford Health Care, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson JT, Pettigrew LE, Teasdale GM. Structured interviews for the Glasgow Outcome Scale and the extended Glasgow Outcome Scale: guidelines for their use. J Neurotrauma. 1998 Aug;15(8):573-85. doi: 10.1089/neu.1998.15.573. PMID 9726257
- [Derived] Schiff ND, Giacino JT, Butson CR, Choi EY, Baker JL, O'Sullivan KP, Janson AP, Bergin M, Bronte-Stewart HM, Chua J, DeGeorge L, Dikmen S, Fogarty A, Gerber LM, Krel M, Maldonado J, Radovan M, Shah SA, Su J, Temkin N, Tourdias T, Victor JD, Waters A, Kolakowsky-Hayner SA, Fins JJ, Machado AG, Rutt BK, Henderson JM. Thalamic deep brain stimulation in traumatic brain injury: a phase 1, randomized feasibility study. Nat Med. 2023 Dec;29(12):3162-3174. doi: 10.1038/s41591-023-02638-4. Epub 2023 Dec 4. PMID 38049620

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Subjects were treated with deep brain stimulation throughout the study, with the exception of a brief, 21 day blinded withdrawal phase that was be undertaken to assess for any possible therapeutic effect.
  Deep brain stimulation: Delivery of continuous, low-voltage electrical pulses to deep portions of the brain via an implantable pacemaker-like device.
Period: Hospital Admission and Surgery (3 Days)
Arm/Group | Treatment
Started | 6
Completed | 6
Not Completed | 0
Period: Post-surgical Washout (65 to 93 Days)
Arm/Group | Treatment
Started | 6
Completed | 5
Not Completed | 1
Not completed — Device explantation | 1
Period: DBS Titration-Optimization (14 Days)
Arm/Group | Treatment
Started | 5
Completed | 5
Not Completed | 0
Period: Unblinded Treatment Phase (90 Days)
Arm/Group | Treatment
Started | 5
Completed | 5
Not Completed | 0
Period: Withdrawal Phase (21 Days)
Arm/Group | Treatment
Started | 3 (2 participants did not participate in the Withdrawal Phase (declined stimulator deactivation) but did proceed to the Continuation Phase.)
Completed | 3
Not Completed | 0
Period: Continuation Phase (6 Months)
Arm/Group | Treatment
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 34 [22 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6
Years since injury [Median (Inter-Quartile Range); unit: years] | 6.5 [3.25 to 9.75]
Years of education [Median (Inter-Quartile Range); unit: years] | 14 [13.25 to 14.00]
Trail-making test, part B [Median (Inter-Quartile Range); unit: seconds] — This test requires the connection of circles marked by numbers and letters in alternating sequence and is considered a benchmark of executive function. The test score is the time required to complete the task in seconds.
  seconds | 116.9 [52.15 to 163.21]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Trail Making Test Part B Time to Completion
Description: The Trail Making Test is a measure of attention, speed and mental flexibility. It also tests spatial organization, visual pursuits, recall, and recognition. Part A requires the individual to draw lines to connect 25 encircled numbers distributed on a page. Part A tests visual scanning, numeric sequencing, and visuomotor speed. Part B is similar except the person must alternate between numbers and letters and is believed to be more difficult and takes longer to complete. Part B tests cognitive demands including visual motor and visual spatial abilities and mental flexibility. Both sections are timed and the score represents the amount of time required to complete the task. Lower scores (shorter times) correspond to a better outcome.
Time Frame: Pre-surgery baseline to treatment phase end (up to 197 days)
Population: Subjects who completed all study assessments through the open label treatment phase
Measure: Median (Inter-Quartile Range); unit: percent change in time
Arm/Group | Treatment
Number analyzed (Participants) | 5
percent change in time | -25.6 [-42.26 to -23.94]

2. Secondary Outcome: Percent Change in Trail Making Test Part A Time to Completion
Description: as for outcome 1
Time Frame: Pre-surgery baseline to treatment phase end (up to 197 days)
Population: Subjects who completed all study assessments through the open label treatment phase
Measure: Median (Inter-Quartile Range); unit: percent change in time
Arm/Group | Treatment
Number analyzed (Participants) | 5
percent change in time | -27.4 [-33.06 to -25.34]

3. Secondary Outcome: Percent Change in Traumatic Brain Injury Quality of Life - Executive Function Short Form (TBI-QOL) Scale Score
Description: The TBI-QOL was developed as a comprehensive patient-reported outcomes (PRO) measurement system specifically for individuals with TBI. It consists of 20 independent calibrated item banks and 2 uncalibrated scales that measure physical, emotional, cognitive, and social aspects of health-related quality of life. We will administer the short form (6-10 questions each) of the TBI-QOL Fatigue, Attention/Concentration, and Executive Function subscales. Executive Function score range: 10-50, higher scores correspond to better executive function.
Time Frame: Pre-surgery baseline to treatment phase end (up to 197 days)
Population: Subjects who completed all study assessments through the open label treatment phase
Measure: Median (Inter-Quartile Range); unit: percent change in score
Arm/Group | Treatment
Number analyzed (Participants) | 5
percent change in score | 28.0 [19.44 to 53.57]

4. Secondary Outcome: Percent Change Traumatic Brain Injury Quality of Life - Attention/Concentration Short Form Scale Score
Description: The TBI-QOL was developed as a comprehensive patient-reported outcomes (PRO) measurement system specifically for individuals with TBI. It consists of 20 independent calibrated item banks and 2 uncalibrated scales that measure physical, emotional, cognitive, and social aspects of health-related quality of life. We will administer the short form (6-10 questions each) of the TBI-QOL Fatigue, Attention/Concentration, and Executive Function subscales. Attention/Concentration score range: 6-30, higher scores correspond to better attention and concentration.
Time Frame: Pre-surgery baseline to treatment phase end (up to 197 days)
Population: Subjects who completed all study assessments through the open label treatment phase
Measure: Median (Inter-Quartile Range); unit: percent change in score
Arm/Group | Treatment
Number analyzed (Participants) | 5
percent change in score | 66.7 [57.85 to 92.86]

5. Secondary Outcome: Percent Change in Traumatic Brain Injury Quality of Life - Fatigue Short Form Scale Score
Description: The TBI-QOL was developed as a comprehensive patient-reported outcomes (PRO) measurement system specifically for individuals with TBI. It consists of 20 independent calibrated item banks and 2 uncalibrated scales that measure physical, emotional, cognitive, and social aspects of health-related quality of life. We will administer the short form (6-10 questions each) of the TBI-QOL Fatigue, Attention/Concentration, and Executive Function subscales. Fatigue score range: 10-50, lower scores correspond to less fatigue.
Time Frame: Pre-surgery baseline to treatment phase end (up to 197 days)
Population: Subjects who completed all study assessments through the open label treatment phase
Measure: Median (Inter-Quartile Range); unit: percent change in score
Arm/Group | Treatment
Number analyzed (Participants) | 5
percent change in score | 2.9 [-20.00 to 5.00]

6. Secondary Outcome: Percent Change in Rivermead Post-Concussion Symptom Questionnaire Scale Score
Description: The Rivermead PCS Questionnaire (RPQ) was originally developed as a measure of severity of symptoms following mild TBI. It consists of 16 post-concussion symptoms including headaches, dizziness, nausea/vomiting, noise sensitivity, sleep disturbance, fatigue, irritability, feeling depressed/tearful, feeling frustrated/ impatient, forgetfulness, poor concentration, taking longer to think, blurred vision, light sensitivity, double vision and restlessness. In the original version of the RPQ, participants are asked to rate the degree (on a scale of 0 to 4) to which a particular symptom has been absent or a mild, moderate or severe problem over the previous 24 hours compared with premorbid levels. Score range: 0-64, lower scores correspond to fewer symptoms
Time Frame: Pre-surgery baseline to treatment phase end (up to 197 days)
Population: Subjects who completed all study assessments through the open label treatment phase
Measure: Median (Inter-Quartile Range); unit: percent change in score
Arm/Group | Treatment
Number analyzed (Participants) | 5
percent change in score | -36.6 [-62.16 to -6.25]

7. Secondary Outcome: Percent Change in Ruff 2 and 7 Automatic Detection Speed Score
Description: The Ruff 2 & 7 Test was developed to measure two aspects of visual attention: sustained attention (ability to maintain consistent performance level over time) and selective attention (ability to select relevant stimuli while ignoring distractors). The test consists of a series of 20 trials of a visual search and cancellation task. The respondent detects and marks through all occurrences of the two target digits: "2" and "7." In the 10 Automatic Detection trials, the target digits are embedded among alphabetical letters that serve as distractors. In the 10 Controlled Search trials, the target digits are embedded among other numbers that serve as distractors. Correct hits and errors are counted for each trial and serve as the basis for scoring the test. Speed scores reflect the total number of correctly identified targets (hits). Score range: 0 to 300, with higher numbers representing more correctly identified targets within the allotted time (5 minutes)
Time Frame: Pre-surgery baseline to treatment phase end (up to 197 days)
Population: Subjects who completed all study assessments through the open label treatment phase
Measure: Median (Inter-Quartile Range); unit: percent change in score
Arm/Group | Treatment
Number analyzed (Participants) | 5
percent change in score | 21.1 [3.87 to 23.17]

8. Secondary Outcome: Percent Change in Ruff 2 and 7 Automatic Detection Accuracy Score
Description: The Ruff 2 & 7 Test was developed to measure two aspects of visual attention: sustained attention (ability to maintain consistent performance level over time) and selective attention (ability to select relevant stimuli while ignoring distractors). The test consists of a series of 20 trials of a visual search and cancellation task. The respondent detects and marks through all occurrences of the two target digits: "2" and "7." In the 10 Automatic Detection trials, the target digits are embedded among alphabetical letters that serve as distractors. In the 10 Controlled Search trials, the target digits are embedded among other numbers that serve as distractors. Correct hits and errors are counted for each trial and serve as the basis for scoring the test. Accuracy scores evaluate the number of targets identified in relation to the number of possible targets (n=300), expressed as a percentage. Higher scores represent higher accuracy of target identification.
Time Frame: Pre-surgery baseline to treatment phase end (up to 197 days)
Population: Subjects who completed all study assessments through the open label treatment phase
Measure: Median (Inter-Quartile Range); unit: percent change in score
Arm/Group | Treatment
Number analyzed (Participants) | 5
percent change in score | 5.2 [1.83 to 7.94]

9. Secondary Outcome: Percent Change in Ruff 2 and 7 Controlled Search Speed Score
Description: as for outcome 7
Time Frame: Pre-surgery baseline to treatment phase end (up to 197 days)
Population: Subjects who completed all study assessments through the open label treatment phase, and who had calculable scores
Measure: Median (Inter-Quartile Range); unit: percent change in score
Arm/Group | Treatment
Number analyzed (Participants) | 4
percent change in score | 17.3 [14.47 to 25.39]

10. Secondary Outcome: Percent Change in Ruff 2 and 7 Controlled Search Accuracy Score
Description: as for outcome 8
Time Frame: Pre-surgery baseline to treatment phase end (up to 197 days)
Population: Subjects who completed all study assessments through the open label treatment phase, and who had calculable scores
Measure: Median (Inter-Quartile Range); unit: percent change in score
Arm/Group | Treatment
Number analyzed (Participants) | 4
percent change in score | 2.7 [1.29 to 5.03]

11. Secondary Outcome: Percent Change in Patient Health Questionnaire - 9 Scale Score.
Description: The Participant Health Questionnaire 9 is a standardized assessment instrument designed to screen, diagnose, monitor, and measure the severity of depression. Score range: 0 to 27, lower scores correspond to better health outcomes.
Time Frame: Pre-surgery baseline to treatment phase end (up to 197 days)
Population: Subjects who completed all study assessments through the open label treatment phase
Measure: Median (Inter-Quartile Range); unit: percent change in score
Arm/Group | Treatment
Number analyzed (Participants) | 5
percent change in score | -41.7 [-80.00 to -30.77]

12. Secondary Outcome: Number of Participants With ≥1 Point Increase in Glasgow Outcome Scale - Extended Scale Score
Description: The Glasgow Outcome Scale Extended (GOS-E) is a measure of disability and handicap intended for use following head injury. The GOS-E subdivides the upper three categories of the original Glasgow Outcome Scale (GOS), severe disability, moderate disability and good recovery, into an eight-category scale: 1 = dead, 2 = vegetative state, 3 = lower severe disability, 4 = upper severe disability, 5 = lower moderate disability, 6 = upper moderate disability, 7 = lower good recovery, and 8 = upper good recovery to provide more detailed assessment of the functional effects of the injury. A structured interview has been developed to standardize assignment of an outcome category (Wilson et al. 1998). Increase of 1 point on this scale represents a meaningful change in health outcome.
Time Frame: Pre-surgery baseline to treatment phase end (up to 197 days)
Population: Subjects who completed all study assessments through the open label treatment phase
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 2

ADVERSE EVENTS:
Time Frame: 1 year (treatment phase plus continuation phase)
Description: Adverse events are presented in a single group because the study was designed to assess any adverse events during the study as a whole, not whether adverse events were associated with any particular study phase.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=6)
Infection of DBS device (Infections and infestations) | 1 (1) — Infection of deep brain stimulator system, requiring removal
Syncope (Nervous system disorders) | 1 (1) — Syncope when standing to urinate
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=6)
Fatigue (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Wound site bleeding (Surgical and medical procedures) | 1 (1) — Scabbing at surgical site with small amount of bleeding
Unintended stimulator deactivation (Product Issues) | 1 (1) — Stimulator de-activated unintentionally (felt to be due to theft detector in store)
Gait disturbance (Nervous system disorders) | 1 (1) — Gait unsteadiness (self limited)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower extremity pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tinnitus (Nervous system disorders) | 1 (1)
Cognitive difficulty (Nervous system disorders) | 1 (1) — Difficulty with planning, organization and word recall
COVID-19 (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT02881151/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/51/NCT02881151/ICF_000.pdf